CLINICAL TRIAL: NCT03820050
Title: FreeStyle LIbre Flash Glucose Monitoring System Pediatric Accuracy Study
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-VAL-18175
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Freestyle LIbre Flash Glucose Monitoring System — System Performance will be characterized with respect to YSI reference venous plasma measurements

SUMMARY:
The purpose of this study is to characterize the Freestyle Libre Flash Glucose Monitoring System in pediatric subjects with respect to YSI reference venous plasma sample measurements.

DETAILED DESCRIPTION:
Up to 250 subjects will be enrolled at up to six (6) clinical research sites in the United States. Subjects will wear two Sensors. Each Sensor will have a paired Reader that will be given to the subject. All Readers will be masked during the study (i.e. subjects will not be able to view glucose results obtained from the Sensor on the Reader screen). Subjects will be asked to perform at least 4 capillary Blood Glucose (BG) tests per day using the primary Reader. Interstitial glucose readings from each Sensor will be obtained with the corresponding Readers immediately following each BG test. Subjects will be instructed to report any problems with the device. Subjects will make three (3), four (4) or five (5) scheduled visits to the clinical study site, including the Enrollment/Screening Visit (Visit 1). Based on the subjects weight, subjects will have up to two (2) in-clinic visits during which intravenous blood draws and YSI reference testing will occur.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between the ages of 4 and 17 years of age at the time of study enrollment.
* Subject must have type 1 or type 2 diabetes.
* Subjects age 11 and older must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily).
* Willing to perform a minimum of 4 finger sticks per day while wearing the sensor in the study.
* Subject and/or guardian must be able to read and understand English.
* For subjects age 6 and older: willing to allow medical personnel to insert an IV catheter in the arm to allow for venous blood flow samples to be obtained per the study protocol.
* For subjects age 11 and older: subject is willing to have their blood sugar manipulated during one or more in-clinic sessions.
* In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
* At the time of enrollment, subject must be available to participate in all study visits.
* Known insulin sensitivity factor (only applicable to subjects age 11 and older).
* Subject's parent, guardian or legally authorized representative must be willing and able to provide written informed consent.
* Subject must be willing and able to provide written signed and dated informed assent when appropriate.

Exclusion Criteria:

* Subject is 18 years of age or older.
* Subject has a history of hypoglycemia unawareness (only applicable to subjects age 11 and older).
* Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
* Subject is known to be pregnant or becomes pregnant during the study (applicable to female subjects only).
* Subject has extensive skin changes/diseases at the proposed application sites that could interfere with device placement or the accuracy of interstitial glucose measurements. Such conditions include, but are not limited to extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, dermatitis herpetiformis, skin lesions, redness, infection or edema.
* Subject has had an episode of severe hypoglycemia requiring intervention from a health care professional(i.e. EMT assistance, emergency room visit, or hospital admission) within the last six (6) months (only applicable to subjects age 11 or older).
* Subject has had an episode of diabetic ketoacidosis (DKA) within the last (3) months (only applicable to subjects age 11 or older).
* Subject is currently participating in another clinical trial.
* Subject has donated blood within 112 days (3.7 months) prior to the beginning of the study activities (only applicable to subjects age 6 and older).
* Subject has both hemoglobin (Hb) and hematocrit levels that are below the normal ranges (only applicable to subjects age 6 and older). The low end of the normal range for Hb is as follows: for males and females aged 6-12 years old it is 11.5 g/dL; for males aged 12-17 it is 13.0 g/dL; for females aged 12-17 it is 12.0 g/dL. The low end of the normal hematocrit for males and females aged 6-12 is 35%; 37% for males aged 12-17 and 36% for females aged 12- 17).
* Subject has X-ray, MRI, CT or diathermy appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
* Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric subjects aged 4-17 with Type 1 or Type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
System Performance | 45 days
  System Performance will be characterized with respect to YSI reference venous plasma measurements

CONTACTS AND LOCATIONS:
Overall Officials: Shridhara Karinka, Ph.D., Study Director — Abbott Diabetes Care
Locations (4):
- United States (4):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alva S, Bailey T, Brazg R, Budiman ES, Castorino K, Christiansen MP, Forlenza G, Kipnes M, Liljenquist DR, Liu H. Accuracy of a 14-Day Factory-Calibrated Continuous Glucose Monitoring System With Advanced Algorithm in Pediatric and Adult Population With Diabetes. J Diabetes Sci Technol. 2022 Jan;16(1):70-77. doi: 10.1177/1932296820958754. Epub 2020 Sep 19. PMID 32954812